CLINICAL TRIAL: NCT06512324
Title: Operation of Brain Stimulation Equipment Under Remote Viewing Effectiveness Registry (OBSERVER)
Brief Title: Operation of Brain Stimulation Equipment Under Remote Viewing Effectiveness Registry
Acronym: OBSERVER
Status: Enrolling by invitation | Type: Observational
Sponsor: Biomedical Discoveries and Neuroscientific Foundations LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: BDNF-001
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Major Depressive Disorder; MDD; Generalized Anxiety Disorder; GAD; Depression; Anxiety
Keywords: Transcranial Magnetic Stimulation; TMS; Noninvasive Brain Stimulation; Accelerated Protocol; Stimulation Parameters; Patient Health Questionnaire; Behavioral Factors; Physiological Factors; Generalized Anxiety Disorder 7-item Scale; PHQ-9; PHQ9; GAD-7; GAD7; Longitudinal Observational Study; Registry; Patient Characteristics; Pharmacological Factors; United States of America; USA, US; Canada; Hamilton Depression Rating Scale; Montgomery-Asberg Depression Rating Scale; Hamilton Anxiety Rating Scale; Generalized Anxiety Disorder 10-item Scale for Adolescents; GAD-10-A, GAD-10A, GAD10, GAD10A; Patient Health Questionnaire for Adolescents; PHQ-9A, PHQ9A
MeSH Terms: conditions — Depressive Disorder, Major; Generalized Anxiety Disorder; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Ampa One TMS System — Transcranial Magnetic Stimulation

SUMMARY:
The goal of this observational study is to record and analyze factors putatively affecting the clinical outcomes among patients undergoing transcranial magnetic stimulation (TMS) treatment for major depressive disorder (MDD) or generalized anxiety disorder (GAD). The main questions it aims to answer are:

1. Which factors have the greatest causal role in mediating the effectiveness of TMS in improving symptoms of depression (and/or anxiety)?
2. Which factors have a minimal causal role in mediating the effectiveness of TMS in improving symptoms of depression (and/or anxiety)?

Participants already undergoing TMS as part of their treatment plan for MDD/GAD answer survey questions about their symptoms before, during, and up to 1 year post-treatment. Factors affecting clinical outcomes such as stimulation parameters, behavioral factors, physiological factors, patient characteristics, and pharmacological factors, are also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Have a primary diagnosis of major depressive disorder (MDD) and/or generalized anxiety disorder (GAD)
* Are receiving outpatient care,
* Voluntarily provide competent consent for treatment,
* Are 12 years of age or older,
* Are able to adhere to the weekly assessment schedule for primary outcome measures,
* Have been assessed by their prescribing physician as suitable candidates for TMS treatment in terms of safety and presenting indication,
* Have consented to undergo a therapeutic course of TMS treatment at one of the participating clinic sites,
* Are able to communicate in the English language.

Exclusion Criteria:

* Have been found to have any contraindication to TMS treatment by their prescribing physician,
* Are considered unsuitable for outpatient care due to illness severity or other factors in the opinion of their prescribing physician,
* Have active suicidal intent or plan,
* Are unable to adhere to or decline participation in the weekly assessment schedule for primary outcome measures,
* Lack the ability to communicate in the English language.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include male, female, and nonbinary patients who are experiencing symptoms of depression and/or anxiety and who have elected to undergo TMS treatment at a participating TMS treatment site, after having been deemed suitable for treatment by their prescribing physician. Participants will have voluntarily chosen to undergo a clinical course of TMS treatment at participating between June 27, 2024, to December 31, 2029. Eligible individuals must be 12 years or older, and participation is limited to those who understand English due to the availability of an English-only informed consent form (ICF).
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2028-08-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
9-item Patient Health Questionnaire (PHQ-9) [or PHQ-9-A if appropriate] | Administered weekly from baseline up to 1 year from the end of treatment.
  The PHQ-9 gauges depressive symptoms through its 9-item brief inventory, efficiently quantifying a spectrum of symptoms, including mood, energy, concentration, sleep, appetite, and suicidality. Widely adopted in outpatient care due to its reliability and validity, the PHQ-9 is a well-established tool in TMS practice, and has shown greater likelihood to detect improvement and less likelihood to miss response or remission among patients undergoing TMS treatment (Leuchter et al. 2023). The PHQ-9-A is the adolescent version of the PHQ-9.
7-item General Anxiety Disorder Questionnaire (GAD-7) [or GAD-10-A if appropriate] | Administered weekly from baseline up to 1 year from the end of treatment.
  The GAD-7, a concise self-report questionnaire evaluating the severity of Generalized Anxiety Disorder (GAD) symptoms, is comprised of seven items. Respondents rate the frequency of experiences over the past two weeks on a Likert scale, resulting in a total score ranging from 0 to 21. The GAD-7 is a streamlined and effective measure, capturing core symptoms such as excessive worrying, restlessness, irritability, muscle tension, and sleep disturbances. It is likewise widely used in real-world TMS practices and registries of TMS outcomes (Sackeim et al. 2020). The GAD-10-A is the adolescent version of the GAD-7.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (HAM-D) [if administered] | Administered weekly from baseline up to 1 year from the end of treatment.
  A clinician-administered 17-item scale assessing neurovegetative, mood and hedonic, cognitive, and other symptom domains, widely used in major studies of TMS in depression (Blumberger et al. 2018).
Montgomery-Asberg Depression Rating Scale (MADRS) [if administered] | Administered weekly from baseline up to 1 year from the end of treatment.
  A 10-item clinician-rated scale assessing emotional, cognitive, and psychomotor aspects of depression, also widely used in TMS research studies (e.g., (O'Reardon et al. 2007; George et al. 2010)).
Hamilton Anxiety Rating Scale (HAM-A) [if administered] | Administered weekly from baseline up to 1 year from the end of treatment.
  A clinician-administered 14-item scale psychological questionnaire used to assess the severity of a person's anxiety; it measures both psychic anxiety and somatic anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Downar, MD PhD FRCPC, Principal Investigator — AMPA Health, Inc.
Locations (2):
- United States (2):
  - Kind Health Group, Encinitas, California
  - Salience Research Institute, Plano, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leuchter MK, Citrenbaum C, Wilson AC, Tibbe TD, Jackson NJ, Krantz DE, Wilke SA, Corlier J, Strouse TB, Hoftman GD, Tadayonnejad R, Koek RJ, Slan AR, Ginder ND, Distler MG, Artin H, Lee JH, Adelekun AE, Leuchter AF. A comparison of self- and observer-rated scales for detecting clinical improvement during repetitive transcranial stimulation (rTMS) treatment of depression. Psychiatry Res. 2023 Dec;330:115608. doi: 10.1016/j.psychres.2023.115608. Epub 2023 Nov 14. PMID 37984281
- [Background] Sackeim HA, Aaronson ST, Carpenter LL, Hutton TM, Mina M, Pages K, Verdoliva S, West WS. Clinical outcomes in a large registry of patients with major depressive disorder treated with Transcranial Magnetic Stimulation. J Affect Disord. 2020 Dec 1;277:65-74. doi: 10.1016/j.jad.2020.08.005. Epub 2020 Aug 7. PMID 32799106
- [Background] Blumberger DM, Vila-Rodriguez F, Thorpe KE, Feffer K, Noda Y, Giacobbe P, Knyahnytska Y, Kennedy SH, Lam RW, Daskalakis ZJ, Downar J. Effectiveness of theta burst versus high-frequency repetitive transcranial magnetic stimulation in patients with depression (THREE-D): a randomised non-inferiority trial. Lancet. 2018 Apr 28;391(10131):1683-1692. doi: 10.1016/S0140-6736(18)30295-2. Epub 2018 Apr 26. PMID 29726344
- [Background] George MS, Lisanby SH, Avery D, McDonald WM, Durkalski V, Pavlicova M, Anderson B, Nahas Z, Bulow P, Zarkowski P, Holtzheimer PE 3rd, Schwartz T, Sackeim HA. Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial. Arch Gen Psychiatry. 2010 May;67(5):507-16. doi: 10.1001/archgenpsychiatry.2010.46. PMID 20439832
- [Background] O'Reardon JP, Solvason HB, Janicak PG, Sampson S, Isenberg KE, Nahas Z, McDonald WM, Avery D, Fitzgerald PB, Loo C, Demitrack MA, George MS, Sackeim HA. Efficacy and safety of transcranial magnetic stimulation in the acute treatment of major depression: a multisite randomized controlled trial. Biol Psychiatry. 2007 Dec 1;62(11):1208-16. doi: 10.1016/j.biopsych.2007.01.018. Epub 2007 Jun 14. PMID 17573044